CLINICAL TRIAL: NCT05351840
Title: An Open-label, Multiple-dose, Fixed-sequence, 3-Period Study to Evaluate the Pharmacokinetic Interactions and Safety in Healthy Volunteers
Brief Title: To Evaluate the Pharmacokinetic Interactions and Safety in Healthy Volunteers
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: JW Pharmaceutical (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Sequential | Masking: None | Purpose: Other
Other Study IDs: JWP-PVA-101
Record Dates: First submitted 2022-04-14; First posted 2022-04-28 (Actual); Last update posted 2022-08-12 (Actual); Status verified 2022-04

CONDITIONS: Healthy

STUDY DESIGN:
Intervention Model Description: open label, multiple dose, Fixed sequence, 3 Period design
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Period I (Experimental): Subject will receive Drug(LivaloV), then take it by oral, once-daily form Day 1 to Day 7
  Interventions: Drug: LivaloV
- Period II (Experimental): Subject will receive Drug(A), then take it by oral, once-daily form Day 14 to Day 23
  Interventions: Drug: A
- Period III (Experimental): Subject will receive Drug(LivaloVA), then take it by oral, once-daily form Day 24 to Day 30
  Interventions: Drug: LivaloVA

INTERVENTIONS:
Drug: LivaloV — Treatment A, Tablet, Oral, QD for 7 Days
  Other Names: Period I
  Arms: Period I
Drug: A — Treatment B, Tablet, Oral, QD for 10 Days
  Other Names: Period II
  Arms: Period II
Drug: LivaloVA — Treatment C, Tablet, Oral, QD for 7 Days
  Other Names: Period III
  Arms: Period III

SUMMARY:
To evaluate and compare the pharmacokinetic interactions and safety of multiple dose of Treatment A and Treatment B alone and in combination

DETAILED DESCRIPTION:
The objective of this study was to evaluate pharmacokinetic characteristics and safety after oral concurrent administration of Treatment A and Treatment B compared to each single administration in Healthy volunteers.

ELIGIBILITY:
Inclusion Criteria:

* Healthy volunteers, aged between 19 to 45 years (both inclusive) at the screening.
* Subjects who are informed of the investigational nature of this study, and voluntarily agree to participate in this study and signs informed consent

Exclusion Criteria:

* Subjects who have a clinically significant past or present medical history of hepato-biliary, renal, gastrointestinal, respiratory, hematologic/neoplastic, endocrine, urologic, psychiatric, musculoskeletal, immunologic, Otorhinolaryngological, and cardiovascular diseases.
* Subjects who have a medical history and/or condition that is considered to be dangerous to take the study drug.

Ages: 19 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 31 (Actual)
Dates: Start 2020-11-02 (Actual); Primary Completion 2020-12-19 (Actual); Study Completion 2021-01-15 (Actual)

PRIMARY OUTCOMES:
The Pharmacokinetics(PK) parameters AUCss,τ | 0~24 hours
  AUCss,τ in a steady-state after multiple-dose (single or combined administration).
The Pharmacokinetics(PK) parameters Css,max | 0~24 hours
  Css,max in a steady-state after multiple-dose (single or combined administration).

CONTACTS AND LOCATIONS:
Overall Officials: Jang Hee Hong, PI, Principal Investigator — Clinical Trial Center, Chungnam National University Hospital
Locations (1):
- Clinical Trial Center, Chungnam National University Hospital, Daejeon, South Korea